CLINICAL TRIAL: NCT02798874
Title: Chinese People's Liberation Army General Hospital
Brief Title: Effects of Ticagrelor on No-reflow in Patients With Acute ST-segment Elevation Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, associate chief physician, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16qgyyq
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Diseases
Keywords: Ticagrelor; No-reflow; Acute ST-segment elevation myocardial; Reperfusion injury; Percutaneous coronary intervention
MeSH Terms: conditions — Cardiovascular Diseases; Reperfusion Injury | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor Group (Experimental): ticagrelor 180 mg 30 min before PCI and 90 mg for 12 months after surgery
  Interventions: Drug: Ticagrelor
- Clopidogrel Group (Active Comparator): Clopidogrel 600 mg 30 min before PCI and 75 mg for 12 months after surgery
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — ticagrelor 180 mg 30 min before PCI and 90 mg for 12 months after surgery
  Arms: Ticagrelor Group
Drug: Clopidogrel — Clopidogrel 600 mg 30 min before PCI and 75 mg for 12 months after surgery
  Arms: Clopidogrel Group

SUMMARY:
The 'no-reflow' phenomenon after a percutaneous coronary intervention (PCI) in patients with acute ST-segment elevation myocardial infarction (STEMI) is a strong predictor of both short- and long-term mortality. Faster antiplatelet activity and increased levels of adenosine provide a theoretical basis for ticagrelor to effectively prevent no-reflow after PCI. We planned to evaluate the effects of ticagrelor on myocardial no-reflow after PCI for STEMI.

DETAILED DESCRIPTION:
Investigators enrolled 240 patients with STEMI who were admitted to the Chinese PLA General Hospital between September 2013 and March 2015. STEMI was defined as typical chest pain lasting N30 min within the previous 12 h, a clear ST-segment elevation of N0.1 mV in ≥2 contiguous electrocardiographic leads, and elevated blood levels of troponin T. We screen high-risk patients through no-reflow risk prediction model， patients were scheduled to undergo diagnostic cardiac angiography or percutaneous coronary interventions. We randomly assigned eligible patients in a 1:1 ratio to receive either ticagrelor 180 mg or clopidogrel 600 mg 30 min before PCI.

The primary efficacy variable was the prevalence of no-reflow assessed immediately post procedure. Secondary efficacy variables were troponin T (TnT), high sensitivity C-reactive protein (hsCRP), interleukin-6 (IL-6), superoxide dismutase (SOD), malondialdehyde (MDA), endothelin-1 (ET-1), and nitric oxide (NO) level

ELIGIBILITY:
Inclusion Criteria:

* patients with STEMI who were admitted to the Chinese PLA General Hospital

Exclusion Criteria:

* 1.unconscious at presentation; 2.had cardiogenic shock, 3.hypoglycemia, 4.diabetic ketoacidosis; 5.had a history of myocardial infarction, stent thrombosis, or renal insufficiency; 6.had previously undergone coronary artery bypass surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the prevalence of no-reflow, | immediately post procedure
  Anterograde coronary flow in the infarct-related artery was graded according to the thrombolysis in myocardial infarction (TIMI) grading system

SECONDARY OUTCOMES:
main cardiovascular events | 90 days
  bleeding, dialysis, myocardial infarction, heart failure and all-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Dai Yun Chen, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Rezkalla SH, Kloner RA. Coronary no-reflow phenomenon: from the experimental laboratory to the cardiac catheterization laboratory. Catheter Cardiovasc Interv. 2008 Dec 1;72(7):950-7. doi: 10.1002/ccd.21715. PMID 19021281
- [Background] Bolognese L, Carrabba N, Parodi G, Santoro GM, Buonamici P, Cerisano G, Antoniucci D. Impact of microvascular dysfunction on left ventricular remodeling and long-term clinical outcome after primary coronary angioplasty for acute myocardial infarction. Circulation. 2004 Mar 9;109(9):1121-6. doi: 10.1161/01.CIR.0000118496.44135.A7. Epub 2004 Feb 16. PMID 14967718
- [Background] Brosh D, Assali AR, Mager A, Porter A, Hasdai D, Teplitsky I, Rechavia E, Fuchs S, Battler A, Kornowski R. Effect of no-reflow during primary percutaneous coronary intervention for acute myocardial infarction on six-month mortality. Am J Cardiol. 2007 Feb 15;99(4):442-5. doi: 10.1016/j.amjcard.2006.08.054. Epub 2006 Dec 20. PMID 17293180
- [Background] Reffelmann T, Kloner RA. The no-reflow phenomenon: A basic mechanism of myocardial ischemia and reperfusion. Basic Res Cardiol. 2006 Sep;101(5):359-72. doi: 10.1007/s00395-006-0615-2. PMID 16915531
- [Background] Wang JW, Chen YD, Wang CH, Yang XC, Zhu XL, Zhou ZQ. Development and validation of a clinical risk score predicting the no-reflow phenomenon in patients treated with primary percutaneous coronary intervention for ST-segment elevation myocardial infarction. Cardiology. 2013;124(3):153-60. doi: 10.1159/000346386. Epub 2013 Mar 8. PMID 23485798
- [Background] Chen Y, Wang C, Yang X, Wang L, Sun Z, Liu H, Chen L. Independent no-reflow predictors in female patients with ST-elevation acute myocardial infarction treated with primary percutaneous coronary intervention. Heart Vessels. 2012 May;27(3):243-9. doi: 10.1007/s00380-011-0144-2. Epub 2011 Apr 28. PMID 21526420
- [Background] Wang J, Chen YD, Zhi G, Xu Y, Chen L, Liu HB, Zhou X, Tian F. Beneficial effect of adenosine on myocardial perfusion in patients treated with primary percutaneous coronary intervention for acute myocardial infarction. Clin Exp Pharmacol Physiol. 2012 Mar;39(3):247-52. doi: 10.1111/j.1440-1681.2012.05668.x. PMID 22214231
- [Background] Teng R, Oliver S, Hayes MA, Butler K. Absorption, distribution, metabolism, and excretion of ticagrelor in healthy subjects. Drug Metab Dispos. 2010 Sep;38(9):1514-21. doi: 10.1124/dmd.110.032250. Epub 2010 Jun 15. PMID 20551239
- [Background] Wittfeldt A, Emanuelsson H, Brandrup-Wognsen G, van Giezen JJ, Jonasson J, Nylander S, Gan LM. Ticagrelor enhances adenosine-induced coronary vasodilatory responses in humans. J Am Coll Cardiol. 2013 Feb 19;61(7):723-7. doi: 10.1016/j.jacc.2012.11.032. Epub 2013 Jan 9. PMID 23312702
- [Background] Steg PG, James S, Harrington RA, Ardissino D, Becker RC, Cannon CP, Emanuelsson H, Finkelstein A, Husted S, Katus H, Kilhamn J, Olofsson S, Storey RF, Weaver WD, Wallentin L; PLATO Study Group. Ticagrelor versus clopidogrel in patients with ST-elevation acute coronary syndromes intended for reperfusion with primary percutaneous coronary intervention: A Platelet Inhibition and Patient Outcomes (PLATO) trial subgroup analysis. Circulation. 2010 Nov 23;122(21):2131-41. doi: 10.1161/CIRCULATIONAHA.109.927582. Epub 2010 Nov 8. PMID 21060072
- [Background] Wang CH, Chen YD, Yang XC, Wang LF, Wang HS, Sun ZJ, Liu HB. A no-reflow prediction model in patients with ST-elevation acute myocardial infarction and primary drug-eluting stenting. Scand Cardiovasc J. 2011 Apr;45(2):98-104. doi: 10.3109/14017431.2011.558209. Epub 2011 Feb 17. PMID 21329416
- [Background] Jogiya R, Kozerke S, Morton G, De Silva K, Redwood S, Perera D, Nagel E, Plein S. Validation of dynamic 3-dimensional whole heart magnetic resonance myocardial perfusion imaging against fractional flow reserve for the detection of significant coronary artery disease. J Am Coll Cardiol. 2012 Aug 21;60(8):756-65. doi: 10.1016/j.jacc.2012.02.075. Epub 2012 Jul 18. PMID 22818072